CLINICAL TRIAL: NCT04289701
Title: The National Hypertension Registry Study of the "Hypertension Prevention and Control Initiative in China" Project
Brief Title: Hypertension Registry of "Hypertension Prevention and Control Initiative in China"
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Jun Cai, Director，Hypertension Center, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: 2019-ZX20
Record Dates: First submitted 2020-02-25; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Hypertension
Keywords: Hypertension; Blood Pressure Control
MeSH Terms: conditions — Hypertension | interventions — Health Services

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hypertension Cohort: Hypertension patients recruited in the "Hypertension Prevention and Control Initiative in China" project.
  Interventions: Other: Health Services for Systematic Hypertension Management

INTERVENTIONS:
Other: Health Services for Systematic Hypertension Management — The systematic hypertension management health services from the "Hypertension prevention and control initiative in China" project. Main services are as follows:
  1. Healthcare provider training and patient education.
  2. Standardized guideline-based hypertension diagnosis, treatment and management recommendation.
  3. Patient-centered, pan-cycle continuous hypertension management via the organizing framework of NMAH and sharing digital platform.
  4. Periodical Patient follow-up via blood pressure monitor-sharing system and in collaboration with other basic local public health programs.
  5. Outcome and performance evaluation quarterly.
  6. Incentives for healthcare organizations and primary healthcare providers, and subsidies to patients.
  7. Certification for "Honorary Hypertension Centers" at county levels and establishment for hypertension clinics at primary care centers.

SUMMARY:
Hypertension is the leading preventable risk factor of cardiovascular disease globally and in China. Unparalleled to remarkable increase of hypertension burden in China, blood pressure(BP) control is inadequate. A political public health project, "Hypertension Prevention and Control Initiative in China(Chronic Disease Demonstration District Construction)", was initiated in October 2019 for explore a feasible and reproducible archetype for hypertension management and to improve the registration, management, treatment and control rates of hypertension in China. The project is designed to consecutively implement health service strategies in 40 pilot counties covering 31 provinces and around 200,000 hypertension patients in mainland China, via the National Medical Alliance for Hypertension(NMAH). The Hypertension Registry study aims to registry, follow up and observe the clinical features, treatment, blood pressure control and outcomes of all hypertension patients managed in the "Hypertension Prevention and Control Initiative in China" project.

DETAILED DESCRIPTION:
Objective: The study aims to investigate the clinical features, treatment, blood pressure control and outcomes of hypertension patients managed in the "Hypertension Prevention and Control Initiative in China" project.

Study Type: A national, multicenter, observational, prospective cohort study.

Study Design: The cardinal contents of this registry study are as follows:

Introduce the Digital Information System and train in completing case report forms.

Collect sociodemographic information, lifestyle behaviors, self-reported personal medical history, BP, anthropometric measurements, medication at registration, laboratory investigations of hypertension patients managed in the "Hypertension Prevention and Control Initiative in China" project. Build a baseline database of hypertension patients.

Gather the follow up information including general, clinical, therapeutic, prognostic data of all recruits at 3-month intervals over 2 years and build up the follow-up database.

Data management, quality control and statistic analysis: Digital Information Platform for data capture, document and cloud computing has been built and the investigators will manage and analyze data in align with key indicators. The investigators have invited professional statistic analysts to assist analyzing data and a third party to supervise data quality.

Ethics: The Ethics Committee of Fuwai Hospital approved this study. Informed consents before patient enrollment are required.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Residing in the local administrative area for at least 6 months.
3. Hypertension：defined as systolic blood pressure (SBP) ≥140 mmHg and/or /diastolic blood pressure (DBP) ≥90 mmHg and/or use of antihypertensive medication within two weeks.
4. Informed consent.

Exclusion Criteria:

1. patients under pregnancy or lactation.
2. patients with severe liver or renal diseases.
3. patients with history of malignant tumor.
4. patients with mental illness that impair their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study recruits patients managed in the "Hypertension Prevention and Control Initiative in China" project. Eligible criteria for the registry study are equal to the inclusion and exclusion criteria for the project. All adult hypertension residents are eligible except for patients cannot be managed at local primary care centers and needing to be transferred for specialist management or residence management.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change for Blood Pressure Control Rate | at 3-month intervals over 24 months
  Change for blood pressure(BP) control rate (number of patients under BP control divided by number of patients registered) from baseline to follow-ups. BP control is defined as follows:
  1. Office BP Control: Office BP controlled to target (Systolic BP<140mmHg and Diastolic BP<90mmHg)
  2. Home BP Control: Home BP controlled to target (Systolic BP<135mmHg and Diastolic BP<85 mmHg)

SECONDARY OUTCOMES:
Change for Systolic Blood Pressure(SBP) | at 3-month intervals over 24 months
  Change for SBP from baseline to follow-ups
Composite Outcome of Cardiovascular Events at 1-year follow-up | 1 year
  A composite of first occurrence of myocardial infarction, stroke (ischemic or hemorrhagic), hospitalization for unstable angina or acute decompensated heart failure, coronary revascularization, atrial fibrillation, or death from cardiovascular causes
Composite Outcome of Cardiovascular Events at 2-year follow-up | 2 years
  A composite of first occurrence of myocardial infarction, stroke (ischemic or hemorrhagic), hospitalization for unstable angina or acute decompensated heart failure, coronary revascularization, atrial fibrillation, or death from cardiovascular causes
Change for Hypertension Treatment Rate | at 3-month intervals over 24 months
  Change for Hypertension Treatment Rate from baseline to follow-ups. Hypertension treatment rate is defined as the number of patients under current antihypertensive medication therapy divided by the number of patients registered.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Cai, MD,PhD, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (11):
- China (11):
  - The First Affliated Hospital of Anhui Medical University, Hefei, Anhui
  - Chinese Academy of Medical Sciences，Fuwai Hospital, Beijing, Beijing Municipality
  - Beijing Shunyi District Hospital, Beijing, Beijing Municipality
  - First affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The second affiliated hospital of Baotou medical college, Baotou, Inner Mongolia
  - The Second Affilated Hospital Of Nanchang University, Nanchang, Jiangxi
  - Yinchuan First People's Hospital, Yinchuan, Ningxia
  - First Affiliated Hospital, Xian Jiaotong University, Xi’an, Shanxi
  - Teda International Cardiovascular Hospital, Tianjin, Tianjin Municipality
  - FuWai YunNan Cardiovascular Hospital, Kunming, Yunnan